CLINICAL TRIAL: NCT02819700
Title: Evaluation and Characterization of Behavioural Disorders and Dementias by the Behavioural Dysexecutive Syndrome Inventory (BDSI)
Acronym: ISDC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI11-PR-GODEFROY-2
Record Dates: First submitted 2016-06-24; First posted 2016-06-30 (Estimated); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Frontotemporal Dementia; Huntington Disease; Alzheimer Disease; Semantic Dementia; Dementia, Vascular
Keywords: behavioural disorders
MeSH Terms: conditions — Frontotemporal Dementia; Huntington Disease; Alzheimer Disease; Dementia, Vascular; Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Behavioral: prevalence of behavioural dysexecutive syndrome — Behavioural Dysexecutive Syndrome Inventory (ISDC)

SUMMARY:
Behavioural disorders are very common right from the initial stage of dementia and contribute to loss of autonomy. Behavioural dysexecutive disorders have a particular status due to their prevalence and their diagnostic importance, as they often constitute the initial symptoms of Frontotemporal Dementia (FTD), Semantic Dementia (SD) and Huntington's disease (HD) and they are classically more frequent in vascular dementia (VaD) than in Alzheimer's disease (AD). The presence of these disorders at the stage of Mild Cognitive Impairment (MCI) has only been partially evaluated and would increase the risk of progression to dementia. These classical data are based on non-standardized assessments and non-validated diagnostic criteria. The Groupe de Reflexion pour l'Evaluation des Fonctions EXécutives (GREFEX) has developed a standardized assessment tool for behavioural dysexecutive disorders, the Behavioural Dysexecutive Syndrome Inventory (BDSI) and has validated diagnostic criteria for this syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Support to the consultation memory for a neurological disease ( frontotemporal dementia , vascular dementia , Alzheimer's disease , mild cognitive disorder, Huntington's disease ( with genetic diagnosis confirmed : number of CAG triplets > 36 symptomatic : UHDRS score ≥5 ) with MMS > 15
* Age 40 to 85 years
* French
* Informing reliable
* Agreeing to participate in the study.

Exclusion Criteria:

* Presence of other disease disturbing behavior ( current depressive syndrome , schizophrenia, psychosis , past psychiatric disorders requiring a stay > 2 days in a specialized environment ) or cognition (mental retardation , illiteracy , respiratory failure, kidney , liver , heart ) or preventing the realization of the tests ( perceptual or motor deficit ) intrecérébrale pacing therapy or stem cell transplant , patient protected ( under supervision or guardianship ) , pregnant and / or breastfeeding and lack of consent

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: French-speaking subjects between the ages of 40 and 85 years with an MMSE score > 15/30, followed for AD or MCI or VaD or FTD or SD or HD will be selected by their neurologist during a routine memory assessment visit.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2013-01-29; Primary Completion 2018-01-28 (Actual); Study Completion 2018-01-28 (Actual)

PRIMARY OUTCOMES:
ISDC (Behavioural Dysexecutive Syndrome Inventory) | Day 0
  Behavioural Dysexecutive Syndrome Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Olivier GODEFROY, MD, PhD, Principal Investigator — CHU Amiens
Locations (2):
- France (2):
  - CHU Amiens, Amiens
  - CHU Strasbourg, Strasbourg